CLINICAL TRIAL: NCT00677092
Title: An Open Label Phase 2 Pilot Study to Determine the Safety, Efficacy and Tolerability of Gleevec (Imatinib Mesylate) in the Treatment of Nephrogenic Systemic Fibrosis
Brief Title: Pilot Study of Imatinib Mesylate to Treat Nephrogenic Systemic Fibrosis
Acronym: GENESYF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jonathan Kay, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-001945
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Nephrogenic Systemic Fibrosis
Keywords: Treatment; Chronic kidney disease; Fibrosing disorders; Imatinib mesylate
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy; Renal Insufficiency, Chronic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate (IM) Treatment (Experimental): Imatinib mesylate 400 milligrams (mg) orally once daily for 4 months. Dosage was reduced to 200 mg if the participant developed gastrointestinal intolerance or alopecia.
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — 400 mg p.o. daily for 4 months. Dosage was reduced to 200 mg if participants develop gastrointestinal intolerance or alopecia.
  Other Names: Gleevec

SUMMARY:
The purpose of this study is to determine the efficacy of imatinib mesylate in reducing cutaneous thickening and tethering in patients with nephrogenic systemic fibrosis (NSF). The study will also work to assess the safety and tolerability of imatinib mesylate in patients with chronic kidney disease and NSF.

DETAILED DESCRIPTION:
Nephrogenic systemic fibrosis (NSF) is a recently described, extremely debilitating and painful condition that affects individuals with renal failure. Recent reports suggest an association between gadolinium exposure during magnetic resonance (MR) studies and the subsequent development of NSF in patients with chronic renal failure. NSF is characterized by rapidly progressive skin hardening, tethering and hyperpigmentation, predominantly on the extremities. Visceral involvement is rare. Skin biopsies of early NSF lesions demonstrate thickened collagen bundles, mucin deposition, angiogenesis and numerous dermal spindle cells that stain with antibodies to cluster of differentiation 34 (CD34) and procollagen. Cutaneous changes of NSF are present in up to 13% of individuals receiving hemodialysis. Among those patients with clinical evidence of NSF, the principle investigator of this protocol has recently reported that NSF is associated with increased early mortality at 24-months.

There is no proven therapy for this devastating disorder. Anecdotal reports have shown modest improvement in joint mobility and decreased skin thickening with extracorporeal photopheresis and pentoxyphylline.

Increased transforming growth factor (TGF)-beta1 messenger ribonucleic acid (mRNA) on immunostaining has been observed in skin, fascia and striated muscle. Imatinib mesylate, a tyrosine kinase inhibitor, prevents TGF-beta-induced stimulation of collagen and extracellular matrix protein synthesis as well as mRNA expression by normal fibroblasts. This observation led the principal investigator to evaluate imatinib mesylate 400 milligrams (mg) orally (p.o.) daily for 1 year in two participants with NSF. The result was significant softening of previously hardened skin with increased mobility of skin that previously had been tethered to the underlying fascia. After one month of imatinib mesylate, one of the two participants had a 20 degree reduction of his knee flexion contractures.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Biopsy-proven NSF
* Ability to give consent

Exclusion Criteria:

* Known sensitivity to imatinib mesylate or to any of its components
* Pregnant or lactating woman
* Bullous dermatologic disease
* Aspartate aminotransferase / alanine aminotransferase (AST/ALT) >3 x upper limit of normal
* Severe congestive heart failure [New York Heart Association (NYHA) Class III or IV]
* Patients who have received Gleevec in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kay, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todd DJ, Kagan A, Chibnik LB, Kay J. Cutaneous changes of nephrogenic systemic fibrosis: predictor of early mortality and association with gadolinium exposure. Arthritis Rheum. 2007 Oct;56(10):3433-41. doi: 10.1002/art.22925. PMID 17907148
- [Background] Kay J, High WA. Imatinib mesylate treatment of nephrogenic systemic fibrosis. Arthritis Rheum. 2008 Aug;58(8):2543-8. doi: 10.1002/art.23696. PMID 18668587
- [Background] Kay J, Czirjak L. Gadolinium and systemic fibrosis: guilt by association. Ann Rheum Dis. 2010 Nov;69(11):1895-7. doi: 10.1136/ard.2010.134791. No abstract available. PMID 20959325
- [Background] Schmidt-Lauber C, Bossaller L, Abujudeh HH, Vladimer GI, Christ A, Fitzgerald KA, Latz E, Gravallese EM, Marshak-Rothstein A, Kay J. Gadolinium-based compounds induce NLRP3-dependent IL-1beta production and peritoneal inflammation. Ann Rheum Dis. 2015 Nov;74(11):2062-9. doi: 10.1136/annrheumdis-2013-204900. Epub 2014 Jun 9. PMID 24914072
- [Background] Todd DJ, Kay J. Gadolinium-Induced Fibrosis. Annu Rev Med. 2016;67:273-91. doi: 10.1146/annurev-med-063014-124936. PMID 26768242

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate Treatment: Imatinib mesylate 400 mg orally once daily for 4 months. Dosage was reduced to 200 mg if participant developed gastrointestinal intolerance or alopecia.
Period: Overall Study
Arm/Group | Imatinib Mesylate Treatment
Started | 12
Received Study Treatment | 11
Completed | 6
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death Prior to Receiving Treatment | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants with available Baseline data.
Groups:
- Imatinib Mesylate Treatment: Imatinib mesylate 400 mg orally once daily for 4 months. Dosage was reduced to 200 mg if the participant developed gastrointestinal intolerance or alopecia.
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in the Modified Rodnan Skin Score (mRSS) to Assess Skin Tethering
Description: The modified Rodnan Skin Score is the accepted clinical measure of scleroderma skin activity. The investigator assessed the thickening of the skin using the modified Rodnan Skin Score through simple palpation on 17 different skin sites in the fingers, hands, forearms, arms, feet, legs, and thighs (bilaterally) and face, chest, and abdomen (singly). Skin thickness was assessed on a scale of 0 to 3; 0 representing normal skin and 3 being severe thickening. The sum of the individual scores can range from 0 (normal) to 51 (severe thickening in all 17 areas). Percentage change is calculated as the Month 4 Score - Baseline Score/Baseline Score * 100. A negative percentage change indicates improvement.
Time Frame: Baseline and Month 4
Population: All enrolled participants with Baseline and Month 4 data available for analysis.
Measure: Mean (Standard Deviation); unit: percentage change in mRSS score
Groups:
- Imatinib Mesylate Treatment: Imatinib mesylate 400 milligrams (mg) orally once daily for 4 months. Dosage was reduced to 200 mg if the participant developed gastrointestinal intolerance or alopecia.
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 6
percentage change in mRSS score | -24 (14)

2. Secondary Outcome: Change From Baseline in Maximal Extension of Elbows and Knees
Time Frame: Baseline and Month 4
Population: PI left institution in 2009; Data collected cannot be associated with specific participants and analyzed for secondary outcome measure.
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Histologic Appearance of Skin Biopsy
Time Frame: Baseline and Month 4
Population: as for outcome 2
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) for Pain
Time Frame: Baseline and Month 4
Population: as for outcome 2
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score
Time Frame: Baseline and Month 4
Population: as for outcome 2
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Score
Time Frame: Baseline and Month 4
Population: as for outcome 2
Arm/Group | Imatinib Mesylate Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Description: PI left institution in 2009; Data collected cannot be associated with specific participants and analyzed for adverse event data entry.
Arm/Group | Imatinib Mesylate Treatment
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
PI left institution in 2009; Data collected cannot be associated with specific participants and analyzed for secondary outcome measure or adverse event data entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No